CLINICAL TRIAL: NCT05643950
Title: Evaluation of the Efficacy and Cost-effectiveness of the T-Control® Catheter Versus the Foley Type Catheter in Patients With Acute Urinary Retention. Randomized Controlled Pilot Clinical Trial
Brief Title: Effectiveness and Cost-effectiveness of the T-Control® Catheter in Patients With Acute Urine Retention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient recruitment by centers
Sponsor: Rethink Medical SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RM-TCONTROL-2022-01; 2022-002862-34 (EudraCT Number)
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Urinary Retention; Catheter-Associated Urinary Tract Infection; Catheter Complications
Keywords: Catheterisation; T-Control; Urinary catheter; Foley catheter
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Masking Description: Data analysis will be blinded to the intervention arm as well as the laboratories that will carry out the analysis of the urine and catheter samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Foley catheter) (Active Comparator): When randomly allocated to this arm, a conventional Foley-type catheter will be inserted during all the study period (2 weeks). At day 14 after inclusion, the patient will be called for a follow-up visit to remove the catheter.
  Interventions: Device: Foley catheter
- T-Control arm (Experimental): When randomly allocated to this arm, the T-Control catheter will be inserted during all the study period (2 weeks). At day 14 after inclusion, the patient will be called for a follow-up visit to remove the catheter.
  Interventions: Device: T-Control catheter

INTERVENTIONS:
Device: Foley catheter — Silicone Foley catheters are transurethral balloon catheters used for the treatment of bladder emptying disorders, as well as for drainage of urine from the urinary tract, continuous fluid irrigation, and/or medication administration. Its use is suitable for a prolonged period of no more than 29 days and is used in Urology, Internal Medicine, Surgery, Obstetrics and Gynaecology Services.
  For this study, conventional Foley-type catheters whose use is approved in Spain for routine use will be used. Silicone Foley catheters, usually available in 2- and 3-way, are made of silicone and consist of a body, drainage funnel, inflation funnel, irrigation funnel (if present, only on 3-way catheters) and balloon valve. The product is sterile and single use.
  Arms: Control arm (Foley catheter)
Device: T-Control catheter — The T-control® catheter is a flexible, sterile silicone tube with an inflatable balloon at the distal tip, a polytetrafluroethylene membrane integrated into its body, and a sliding fluid control valve. The valve, built into the catheter, provides additional functions to the catheter, such as turning urine flow on and off after insertion (functions currently provided by accessories such as caps or valves) and controlling urination during the insertion process (function that is not provided by any other device). In this way, accidental loss of urine can be avoided from the first moment of use until its withdrawal. Additionally, it has a safety cap that reduces the possibility of accidental movements of the valve before use or during transport and fixing. The design has been developed in such a way that, once inserted, it facilitates autonomous use even for the elderly or patients with limited manual dexterity. The device is sterile and single use, like any conventional Foley catheter.
  Arms: T-Control arm

SUMMARY:
The general purpose of this study is to assess the preliminary effectiveness and cost-effectiveness of the T-Control® catheter versus the Foley type catheter in patients with Acute Urine Retention.

DETAILED DESCRIPTION:
Potential participants will be identified by the team of healthcare professionals of the emergency department according to the inclusion and exclusion criteria of the study. If the patient meets the criteria, the emergency department team will be able to refer patients directly to the urology department, where the investigator or research assistant will again check the inclusion and exclusion criteria, will invite the patient or their relative/caregiver (if necessary) to participate in the study and will request their informed consent. The catheter insertion will be carried out by the research staff after the inclusion and randomisation of the participants.

After catheter insertion, participants and their family, friends, or other informal caregivers will receive information about wearing an indwelling urinary catheter and specific information to randomly inserted, standard Foley, or T-Control® catheters. Standard catheter care is permitted during the trial both managed by the participants and participants' caregivers. Additionally, participants will receive an incident diary in which participants can record any type of incident during the bladder catheterisation period. Two weeks after indwelling bladder catheter insertion, participants will be contacted by urology outpatients for a follow-up visit, during which the study catheter will be removed.

Finally, within a maximum period of two weeks after the follow-up visit, the participants will be invited to participate in an interview to assess the quality of life perceived by the participants during the study

ELIGIBILITY:
Inclusion Criteria:

* Males with Acute Urine Retention
* Equal or over 50 years of age
* Absence of symptoms of infection on the inclusion day
* Not having been previously catheterized on the day of inclusion
* Indication of bladder catheterization for 2 weeks
* Maintained cognitive and physical capacity for self-monitoring the catheter valve
* Signed consent agreement

Exclusion Criteria:

* Current or recent urinary tract infection in the last 2 weeks
* Use of current treatment/antibiotic in the last 2 weeks
* Immunocompromised patients (diagnosed with advance cancer, Acquired Immunodeficiency Syndrome,...)
* Catheter insertion requiring more than 1 attempt
* Overactive bladder
* Patients with bilateral obstructive uropathy

Ages: 50 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Magnitude of infections | Day 14 after inclusion (follow-up visit)
  The magnitude of infection will be obtained from the analysis of urine culture samples taken from participants

SECONDARY OUTCOMES:
Rate of symptomatic and asymptomatic infections | Day 14 after inclusion (follow-up visit)
  The magnitude of infection obtained from the urine samples will be classified according to the following criteria: Symptomatic infection: the presence of pathogenic microorganisms in amounts greater or equal to 1,000 CFU/mL accompanied with symptoms will determine the existence of the infection; Asymptomatic infection: in the absence of infection symptoms, a determination of microorganisms greater than or equal to 100,000 CFU/mL will indicate asymptomatic infection. In addition to the presence or absence of infections to assess their rate, this variable will also be collected using the outcome measure "infection-free days" (with a maximum possible value of 14 days).
Self-perceived health-related quality of life (HRQoL) | Day 14 after inclusion (follow-up visit)
  The following instruments are administered to participants: EuroQol-5 Dimensions-5 Levels (this is a generic health-related quality of life questionnaire that evaluates five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The questionnaire also includes a visual analogue scale) and a Catheter-related Quality of Life questionnaire (Rethink Medical developed a specific instrument created in the context of this project based on the experience of our previous studies. The questionnaire consists of questions that collect data on the prescription of the bladder catheter and on the accessories used (collection bag, plugs or others), questions related to acceptability, usability and satisfaction in relation to the catheter and the accessories used, adverse events and changes in habits in relation to the catheter and emotions perceived at the beginning and during the use of the bladder catheter).
Indication of antibiotic treatments | Day 14 after inclusion (follow-up visit)
  The antibiotic that has been administered associated with the use of the catheter will be recorded along with the dose and treatment time.
Determination of the biofilm formed in the catheters | Day 14 after inclusion (follow-up visit)
  The catheter removed will be sent to the laboratory and it will be cultured to assess the presence or absence of biofilm. The microorganisms forming the biofilm will be quantified as colony-forming units/catheter pieces. Also, these microorganisms will be identified in order to establish statistical relationships with those identified in the urine cultures.
Number of adverse events related to catheterization | Day 14 after inclusion (follow-up visit)
  The type and number of adverse events will be recorded: accidental disconnection of the catheter, obstruction, pain, loss of urine per catheter, haematuria and accidental spills caused by the professional during the moment of insertion.
Total costs of each type of catheterization (cost-effectiveness) per quality-adjusted life year (QALY) of catheterized participants | Close-out of the study
  The costs derived from the catheterization, such as the consumption of consumable materials and resources, diagnostic tests (urine cultures and catheter cultures and biofilm analysis) will be collected. The budgetary impact derived from the incorporation of T-Control® into the service portfolio of Spanish hospitals will be included. The main outcome measure will be the incremental cost per quality-adjusted life year (QALY) gained, a generic health measure that combines information on life expectancy with the patient's quality of life, the latter measured through the EuroQoL-5 Dimensions-5 Levels instrument. The perspective of the analysis will be that of the hospital, in which only direct healthcare costs will be included.
Level of satisfaction and workload of health professionals. | Close-out of the study
  The following instruments are administered to health professionals: National Aeronautics and Space Administration - Task Load Index (The questionnaire evaluates 6 dimensions allowing to rate them on a 1 to 10 scale) and Health professional satisfaction questionnaire (questionnaire specifically developed to quantitatively measure satisfaction with the devices used. This questionnaire includes a first section with 12 statements regarding the catheter insertion process. The second section is intended for health professionals to make a comparison between both devices through 11 statements. Finally, the questionnaire consists of a free section in which health professionals can write any comments or suggestions).
Acceptability of the T-Control® device | Day 14 after inclusion (follow-up visit)
  Patient experience framed in the trajectory of the disease, identifying the preferences and needs for training and information for the use of the device and possible future improvements for the T-Control® device. A subgroup of participants will be selected by means of an intentional theoretical sampling seeking the maximum variability in terms of age and presence of infection. This selection will be made until information saturation is achieved, which is estimated between 10 and 20 participants. For data collection, the technique of in-depth interviews will be used using a semi-structured script. The interviews will be audio recorded and transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vera, Dr., Principal Investigator — Hospital Universitario Insular de Gran Canaria; Adrián Amador, Dr., Principal Investigator — University Hospital of the Nuestra Señora de Candelaria
Locations (2):
- Spain (2):
  - Complejo Hospitalario Universitario Insular Materno-Infantil de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife

IPD SHARING:
Plan to Share IPD: Yes
The requests for participant-level data and/or statistical code can be made in writing to info@rethinkmedical.es. The final trial dataset generated and/or analysed during the study may be available on reasonable request to the research coordinator and Sponsor.
Supporting Information: Study Protocol
Time Frame: Starting 2 months after publication.
Access Criteria: Review requests and criteria for reviewing requests will be carried out by the Principal Investigators and Sponsor.